CLINICAL TRIAL: NCT00269581
Title: Headstrong Intervention for Recurrent Pediatric Headache
Brief Title: Headstrong Intervention for Pediatric Headache
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Michael Rapoff, Ph.D. (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Michael Rapoff, Ph.D., Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9578; NS46641
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Headaches
Keywords: migraine; tension headaches; chronic daily headaches
MeSH Terms: conditions — Headache Disorders; Migraine Disorders; Tension-Type Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): Educational CD-Rom
  Interventions: Other: Educational CD-rom
- 2 (Experimental): Headstrong CD-rom
  Interventions: Other: Headstrong CD-rom

INTERVENTIONS:
Other: Educational CD-rom — Educational CD-Rom
  Arms: 1
Other: Headstrong CD-rom — Headstrong CD-rom
  Arms: 2

SUMMARY:
Purpose of this study is to determine if a CD-ROM computer program (called "Headstrong") is effective in helping children cope with chronic headaches.

DETAILED DESCRIPTION:
Children, 7-12 years, with recurrent headaches are randomly assigned to an educational CD-ROM program or the Headstrong CD-ROM program. We anticipate that those assigned to the active (Headstrong) program group will have significantly greater reductions in headache frequency, duration, and severity and improvements in mood and quality of life.

ELIGIBILITY:
Inclusion criteria:

* 7-12 years of age
* having recurrent, intermittent, nonmalignant headaches occurring on an average of at least once per week by parental or child report and separated by symptom-free periods
* having a diagnosis by a nurse practitioner, pediatrician, or pediatric neurologist of migraine, muscle-contraction, or chronic daily headaches

Exclusion criteria:

* their medical history and/or neurological exam suggests that headaches are secondary to another physical or developmental condition
* their parents report they have been diagnosed with a mental health condition or they are receiving concurrent psychotherapy
* their baseline headache diaries indicate an average headache frequency of less than one per week

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2004-08; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Pain, mood, and stress self-rating scales | Baseline, Immediate Post-Treatment and 3, 6 and 12 Month Follow-Up

SECONDARY OUTCOMES:
Quality of life | Baseline, Immediate Post-Treatment and 3, 6 and 12 Month Follow-Up
Headache-related disability | Baseline, Immediate Post-Treatment and 3, 6 and 12 Month Follow-Up

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rapoff, PhD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Children's Mercy Hospital Kansas City, Kansas City, Missouri